CLINICAL TRIAL: NCT02576028
Title: Fascial Manipulation® Associated With Standard Care Versus Standard Post-surgical Care for Total Hip Arthroplasty: a Randomized Controlled Trial.
Brief Title: Fascial Manipulation® Associated With Standard Care Versus Standard Post-surgical Care for Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Bolognini di Seriate Bergamo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1173-0402
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Arthritis
Keywords: Total Hip Replacement; Manipulation Therapy
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard treathment (Other): two sessions of 45 minutes of active exercises for 10 days
  Interventions: Other: standard active exercises
- FM associated to standard treathment (Experimental): the same intervention of CG except on days 2 and 7 where one session treatment was replaced with a FM treatment.
  Interventions: Other: Fascial Manipulation® (FM); Other: standard active exercises

INTERVENTIONS:
Other: Fascial Manipulation® (FM) — Fascial Manipulation® (FM) is a manual therapy that focus on the deep muscular fascia. This technique considers the fascia as a three-dimensional continuum. The mainstay of this manual technique lies in the identification of specific localised areas of the fascia, defined Center of Coordination (CC), where the gliding of the subcutis should be preserved to avoid biomechanical in-coordination of the surrounding muscles. The method is performed by applying a deep friction over the CCs that result more altered at the clinical palpation
  Arms: FM associated to standard treathment
Other: standard active exercises — two sessions of 45 minutes of active exercises

SUMMARY:
Post-surgical physiotherapy programs following to total hip arthroplasty (THA) show important differences between types and numbers of treatment sessions. Objectives are to investigate effectiveness of Fascial Manipulation when associated to a standard protocol of care.

DETAILED DESCRIPTION:
Background. Post-surgical physiotherapy programs following to total hip arthroplasty (THA) show important differences between types and numbers of treatment sessions. Objectives are to investigate effectiveness of Fascial Manipulation when associated to a standard protocol of care.

Methods. Fifty-one subjects operated with THA were randomized into two groups, both followed a standard protocol of care where two sessions were replaced with Fascial Manipulation in the study group. Functional outcomes measures collected before and after treatment and at the end of the rehabilitation program included Harris Hip Score, Time Up and Go test, articular range of motion and verbal numerical scale.

ELIGIBILITY:
Inclusion Criteria:

* first THA surgery,
* posterior-lateral access,
* onset of pain of maximum 2 years

Exclusion Criteria:

* patients with previous hip or knee prosthesis,
* congenital hip dysplasia,
* revision THA,
* elective THA secondary to trauma,
* real leg-length discrepancy (≥1.5cm),
* cognitive impairment,
* concomitant rheumatic pathology in acute phase,
* serious comorbidities including cardiac,
* respiratory and/or neuromuscular pathologies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
change of pain during movement | change from before and after the 2nd day treatment, change from before and after the 7nd day treatment, change from 2nd and 10th day (end of study)
  value of pain during a specific movement , measured with Visual Numeric Scale (VNS) scale

SECONDARY OUTCOMES:
Range of motion (ROM) | before and after the 2nd day treatment, before and after the 7nd day treatment, 10th day (end of study)
  hip ROM amplitude, measured with bobble inclinometer
Harris Hip Score | before and after the 2nd day treatment, before and after the 7nd day treatment, 10th day (end of study)
  Functional outcome
Timed up and Go test (TuG) | before and after the 2nd day treatment, before and after the 7nd day treatment, 10th day (end of study)
  functional test for stand up and walk speed

REFERENCES:
- [Derived] Busato M, Quagliati C, Magri L, Filippi A, Sanna A, Branchini M, Marchand AM, Stecco A. Fascial Manipulation Associated With Standard Care Compared to Only Standard Postsurgical Care for Total Hip Arthroplasty: A Randomized Controlled Trial. PM R. 2016 Dec;8(12):1142-1150. doi: 10.1016/j.pmrj.2016.04.007. Epub 2016 May 19. PMID 27210234